CLINICAL TRIAL: NCT04949334
Title: Effects of Respiratory Muscle Training in Patients With Acute Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Chen ruey, Assistant professor, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202009012
Record Dates: First submitted 2021-02-04; First posted 2021-07-02 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Stroke, Ischemic
Keywords: Stroke; Respiratory muscle training; Respiratory function
MeSH Terms: conditions — Ischemic Stroke; Stroke; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dofin Breathing Strength Builder (Experimental): Usual post stroke care and respiratory muscle training
  Interventions: Device: Dofin Breathing Strength Builder
- Usual post stroke care (No Intervention): Usual post stroke care

INTERVENTIONS:
Device: Dofin Breathing Strength Builder — If the patient's condition is stable, respiratory muscle training will be performed under Dofin Breathing Strength Builder 7 days after stroke. The patient will receive respiratory muscle training by repetition of 30 times, two courses per day, x 7 days, for three weeks.
  The initial load was set at 30% of the participants' maximal baseline strength and increased weekly at intervals of 2 cmH2O.
  Arms: Dofin Breathing Strength Builder

SUMMARY:
After acute ischemic stroke, the muscle strength of the limbs of the patients will decrease. Moreover, the respiratory muscles may also be affected. The respiratory muscle training may improve the respiratory recovery and prevent pulmonary complication.

DETAILED DESCRIPTION:
After acute ischemic stroke, the muscle strength of the limbs of the patients will decrease. Moreover, the respiratory muscles may also be affected. The worsening of the respiratory function is weakened and lung function declines, leading to dysfunction of expectoration and swallowing, and increasing the incidence of pneumonia after stroke. In addition, it will also lead to a decline in activity ability, which in turn affects the quality of life. The respiratory muscle training may improve the respiratory recovery and prevent pulmonary complication.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic stroke diagnosed by MRI
2. Age over 20 years old
3. No worsening of stroke or second stroke this time

Exclusion Criteria:

1. Unable to understand instructions normally, or communication difficulties
2. Patients with endotracheal tube or tracheostomy
3. Angina in recent 3 months, myocardial infarction, heart failure
4. Patients with asthma or chronic obstructive pulmonary disease, spontaneous pneumothorax, and ongoing pneumonia
5. Patients with untreated hernias
6. Pregnant
7. Ongoing fever (body temperature>38.5°C)
8. Poor hypertension control (higher than 170/100 mmHg three days before intervention)
9. Patients who have had cerebral hemorrhage or aneurysm

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle function-1.1 | Baseline
  MEP (maximal expiratory pressure)
Respiratory muscle function-1.2 | Within one week after training
  MEP (maximal expiratory pressure)
Respiratory muscle function-1.3 | Twelve weeks after training
  MEP (maximal expiratory pressure)
Respiratory muscle function-2.1 | Baseline
  MIP (maximal inspiratory pressure)
Respiratory muscle function-2.2 | Within one week after training
  MIP (maximal inspiratory pressure)
Respiratory muscle function-2.3 | Twelve weeks after training
  MIP (maximal inspiratory pressure)

SECONDARY OUTCOMES:
Dyspnea.1 | Baseline
  Dyspnea assessed by Modified Borg Dyspnea Scale (MBS). MBS can go from 0-10, 10 is the more severe condition.
Dyspnea.2 | Within one week after training
  Dyspnea assessed by Modified Borg Dyspnea Scale (MBS). MBS can go from 0-10, 10 is the more severe condition.
Dyspnea.3 | Twelve weeks after training
  Dyspnea assessed by Modified Borg Dyspnea Scale (MBS). MBS can go from 0-10, 10 is the more severe condition.
Exercise tolerance.1 | Baseline
  Exercise tolerance assessed by six-minute walk test (6MWT).
Exercise tolerance.2 | Within one week after training
  Exercise tolerance assessed by six-minute walk test (6MWT).
Exercise tolerance.3 | Twelve weeks after training
  Exercise tolerance assessed by six-minute walk test (6MWT).
Body composition.1 | Baseline
  Body composition including body fat and muscle mass measured by multi frequency segmental body composition analyzer (TANITA).
Body composition.2 | Within one week after training
  Body composition including body fat and muscle mass measured by multi frequency segmental body composition analyzer (TANITA).
Body composition.3 | Twelve weeks after training
  Body composition including body fat and muscle mass measured by multi frequency segmental body composition analyzer (TANITA).
Life quality.1 | Baseline
  Quality of life assessed by Short-form 12 (SF-12). SF-12 can go from 0-100, 100 is the better life quality.
Life quality.2 | Within one week after training
  Quality of life assessed by Short-form 12 (SF-12). SF-12 can go from 0-100, 100 is the better life quality.
Life quality.3 | Twelve weeks after training
  Quality of life assessed by Short-form 12 (SF-12). SF-12 can go from 0-100, 100 is the better life quality.
Swallowing.1 | Baseline
  Swallowing function assessed by the Functional Oral Intake Scale (FOIS). The score can go from 1-7, 7 is the better oral intake condition.
Swallowing.2 | Within one week after training
  Swallowing function assessed by the Functional Oral Intake Scale (FOIS). The score can go from 1-7, 7 is the better oral intake condition.
Swallowing.3 | Twelve weeks after training
  Swallowing function assessed by the Functional Oral Intake Scale (FOIS). The score can go from 1-7, 7 is the better oral intake condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Shuang Ho Hospital, Taipei Medical University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes